CLINICAL TRIAL: NCT02518854
Title: Identifying Biomarkers and Cardiovascular Risk Factors in Childhood Metabolic Syndrome
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tain, You-Lin, Dr., Chang Gung Memorial Hospital
Other Study IDs: 104-1970A3
Record Dates: First submitted 2015-08-04; First posted 2015-08-10 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Metabolic Syndrome; Cardiovascular Disease
MeSH Terms: conditions — Metabolic Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study: children aged 6-18 years with pre-metabolic syndrome
- control: children aged 6-18 years without pre-metabolic syndrome

SUMMARY:
Metabolic syndrome (MetS) is highly prevalent all over the world. MetS is largely under-diagnosed in children and adolescents. Obesity and hypertension are two important requirements for criteria of MetS. With early detection and early intervention of MetS in children and adolescents will enable better care to reduce the heavy burden of health care all over the world.

Investigators intend to recruit 150 children and adolescents age 6 to 18 yr with overweight/obesity or prehypertension/hypertension and 50 normal age-matched controls to reach the following research goals:

1) To identify biomarkers as risk factors; 2) To characterize that impact of vascular assessment in preMetS children; and 3) To examine the relationship among biomarkers, vascular assessment parameters, and metabolic phenotypes.

DETAILED DESCRIPTION:
Metabolic syndrome (MetS) is highly prevalent all over the world, including Taiwan. So far, there is still no standard definition of MetS for use in pediatric population. Thus MetS is largely under-diagnosed in children and adolescents. Obesity and hypertension are two important requirements for criteria of MetS. With early detection and early intervention of MetS in children and adolescents will enable better care to reduce the heavy burden of health care all over the world.

MetS might originate from early life, namely developmental programming. Cardiovascular disease (CVD) is the most common comorbidity of MetS. Therefore identification of biomarkers for detecting children with high-risk to develop CVD and MetS progression is our priority. Investigators' previous studies identified some biomarkers from a variety of programming models, including asymmetric dimethylarginine (ADMA, a nitric oxide synthase inhibitor), β-trace protein (BTP, also known as lipocalin-type prostaglandin D synthase), and adiponectin. Thus, in the current study, ADMA profile, BTP, and adiponectin will be studied in children and adolescents with pre-MetS to explore their role as biomarkers to predict MetS and CVD progression.

In childhood, assessment of CVD relies on endothelial function and arterial stiffness, as CV events are extremely rare. Thus, in this study investigators intend to perform a global vascular assessment (to determine endothelial function and arterial stiffness) in children with pre-MetS including 24hr ABPM, measure of pulse wave velocity (PWV) and ambulatory arterial stiffness index (AASI) to detect arterial stiffness, detection of flow mediated dilatation (FMD), and biomarkers. Investigators also intend to examine the correlation between biomarkers and these measured vascular parameters in children with preMetS.

Therefore, investigators will recruit 150 children and adolescents age 6 to 18 yr with overweight/obesity or prehypertension/hypertension and 50 normal age-matched controls to reach the following research goals:

1) To identify biomarkers as risk factors; 2) To characterize that impact of vascular assessment in preMetS children; and 3) To examine the relationship among biomarkers, vascular assessment parameters, and metabolic phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* children with ≧ one of the following criteria of metabolic syndrome

  1. weist circumstance ≧90th percentile
  2. TG≧150 mg/dL
  3. HDL<40 mg/dL
  4. BP>≧90th percentile
  5. A.C. glucose>100 mg/dL or T2D
* Volunteer

Exclusion Criteria:

* inability to complete study procedures
* pregnancy
* malignancy.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 6-18 years visit pediatric nephrology clinic during study period
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Asymmetric dimethylarginine (ADMA) | At the time of enrollment
  Differences of ADMA level (μM) in children with pre-Metabolic syndrome vs. control.

SECONDARY OUTCOMES:
Adiponectin | At the time of enrollment
  Differences of adiponectin level (μg/mL) in children with pre-Metabolic syndrome vs. control.
β-trace protein (BTP) | At the time of enrollment
  Differences of BTP level (mg/dL) in children with pre-Metabolic syndrome vs. control.
Flow-mediated dilation (FMD) | At the time of enrollment
  Differences of FMD (%) in children with pre-Metabolic syndrome vs. control.
Pulse wave velocity (PWV) | At the time of enrollment
  Differences of PWV (m/s) in children with pre-Metabolic syndrome vs. control.
Ambulatory arterial stiffness index (AASI) | At the time of enrollment
  Differences of AASI (unit) in children with pre-Metabolic syndrome vs. control.

CONTACTS AND LOCATIONS:
Overall Officials: You-Lin Tain, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan